CLINICAL TRIAL: NCT03422601
Title: Prognostic Value of the Immunoscore® Colon Test for Disease Free Survival Stratification in Stage III Patients Under Oxaliplatin Treatment: an Ancillary Study of IDEA France Study
Brief Title: Prognostic Value of the Immunoscore® Colon Test for Disease Free Survival Stratification in Stage III Patients Under Oxaliplatin Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: HalioDx (Industry); Methodology and quality of life unit in oncology, University hospital of Besancon (Unknown)
Responsible Party: Sponsor
Other Study IDs: IDEA ancillary study
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer; Stage III Colon Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissues: colon carcinoma and adjacent non-tumor tissues collected in formalin fixed paraffin embedded blocks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3 months treatment: FOLFOX or CAPOX
  Interventions: Diagnostic Test: Immunoscore test
- 6 months treatment: FOLFOX or CAPOX
  Interventions: Diagnostic Test: Immunoscore test

INTERVENTIONS:
Diagnostic Test: Immunoscore test — To identify patients with high risk (IS 0-1) of relapse or death under oxaliplatin-based adjuvant therapy.

SUMMARY:
The primary objective is to validate that the Immunoscore® test (IS0 to IS4) is able to identify patients with high risk (IS 0-1) of relapse or death whichever occurs first among Stage III patients under oxaliplatin-based adjuvant therapy.

Then the prognostic value of Immunoscore® Colon to predict disease free survival (DFS) will be assessed in Stage III patients under Oxaliplatin treatment in each arm of the IDEA trial (6- months and 3-months treatment).

Finally, the additive value of the Immunoscore® test to stratify the DFS will be evaluated among standard clinical and biological parameters and tumor features.

DETAILED DESCRIPTION:
Adult patients of both genders who have underwent surgical resection of stage III colon carcinoma and randomised to receive a 6-month or 3-month adjuvant therapy with modified FOLFOX 6 or CAPOX in the IDEA France trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient and tumor characteristics; 3-year clinical Follow-Up
* Data regarding other markers (eg. MSI)
* FFPE blocks available, including core tumor + invasive margin regions

Exclusion Criteria:

• Bouin fixative

Sample type:

• adjacent FFPE slices (4 μm each) per case (although only one slide is required for CD3 and one for CD8, with center of tumor (CT) and the invasive margin(IM) cut from FFPE blocks no more than 4 months before the Immunoscore® testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient of both genders who have underwent surgical resection of stage III colon carcinoma
Sampling Method: Probability Sample
Enrollment: 1122 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 3 years
  DFS is defined as the time from randomization to relapse or death, whichever occurred first. Secondary colon cancers are regarded as DFS events, whereas non-colon tumors are to be disregarded in the analysis. Patients with no defined events observed during the follow-up will be censored at the date of last disease evaluation which showed no evidence of relapse, or secondary primary colon cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry ANDRE, MD, Study Director — Hôpital Saint Antoine
Locations (1):
- Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pages F, Andre T, Taieb J, Vernerey D, Henriques J, Borg C, Marliot F, Ben Jannet R, Louvet C, Mineur L, Bennouna J, Desrame J, Faroux R, Kirilovsky A, Duval A, Laurent-Puig P, Svrcek M, Hermitte F, Catteau A, Galon J, Emile JF. Prognostic and predictive value of the Immunoscore in stage III colon cancer patients treated with oxaliplatin in the prospective IDEA France PRODIGE-GERCOR cohort study. Ann Oncol. 2020 Jul;31(7):921-929. doi: 10.1016/j.annonc.2020.03.310. Epub 2020 Apr 12. PMID 32294529